CLINICAL TRIAL: NCT06030557
Title: PrEPared-RN, CAN Nurse-Led Management of High-risk Patients for Pre-Exposure
Brief Title: PrEPared-RN, CAN Nurse-Led Management of High-risk Patients for Pre-Exposure Prophylaxis (PrEP)
Acronym: Prep-RN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CAN Community Health (Other)
Responsible Party: Sponsor
Other Study IDs: IN-US-412-6439
Record Dates: First submitted 2023-02-02; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-02

CONDITIONS: Hiv Prevention; Pre-Exposure Prophylaxis (PrEP)
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Truvada — Participants will receive either Truvada or Descovy (based on prescription guidelines).
  Other Names: Descovy

SUMMARY:
During the initial encounter, the nurses will complete program enrollment forms (consents and disclosures as approved by IRB), medical history, and risk assessment. If needed, the RN will facilitate a 4th generation rapid HIV test or draw HIV serology. A general review of systems, focused physical exam with emphasis on sexually transmitted infections and signs of seroconversion is provided, including identifying signs of genitourinary infection.

The nurse will order labs per standing order and performs blood draw. Pre-test and Post-test counseling with HIV and STI testing is provided at this time. Upon receipt of a negative HIV rapid or serology test, PrEP-RN provides a 7-14 day supply of samples with a 30-day prescription of FTC/TDF (Truvada) or a 30-day prescription of FTC/TAF (Descovy) per standing order.

At each follow-up visit, client's self-efficacy, attitudes/beliefs about PrEP, general health indicators, and social determinants of health, such as access to transportation and housing status, are recorded. Process evaluation will be performed to determine relationships of these variables and PrEP adherence, implementation (12 months), and continuation/dissemination (year 2) phases of the study.

DETAILED DESCRIPTION:
The following study design is an alternative to the existing protocol at CAN clinics. The point of care will be RN-led, as opposed to the Provider. The Provider will still retain safety and protocol oversight, but the RN will make the clinical decisions. Findings of this study will demonstrate the relative efficacy of the nurse-led PrEP services in comparison to the traditional provider-led services.

During the initial three months of the study period, CAN will hire and train two registered nurses with licensure in the State of Florida. These nurses will work with Shannon DiPalmo, MSW, CANs Vice President for Community Engagement and other staff to identify community, faith-based organizations, and colleges who serve the priority populations. CAN will establish memoranda of agreement with these organization to allow regular visits by nurses to meet with participants in safe, private spaces where PrEP services can be provided in person or through telehealth.

When these relationships are established, the RNs will work with the partner to schedule PrEP encounters. CAN plans to enroll a minimum of 210 study participants at a minimum of six different locations.

During the initial encounter, the nurses will complete program enrollment forms (consents and disclosures as approved by IRB), medical history, and risk assessment. If needed, the RN will facilitate a 4th generation rapid HIV test or draw HIV serology. A general review of systems, focused physical exam with emphasis on sexually transmitted infections and signs of seroconversion is provided, including identifying signs of genitourinary infection (e.g., discharge, lesions, or pain), rectal infection (anal pain, tenesmus, or discharge). This exam also includes an inspection of the oral mucosa for signs of primary or secondary syphilis. The nurse will order labs per standing order and performs blood draw. Pre-test and Post-test counseling with HIV and STI testing is provided at this time. Upon receipt of a negative HIV rapid or serology test, PrEP-RN provides a 7-14 day supply of samples with a 30-day prescription of FTC/TDF (Truvada) or a 30-day prescription of FTC/TAF (Descovy) per standing order. The RN schedules a 2-week follow-up phone call with the patient and a 4-week follow-up and lab-draw visit. At the 2-week follow-up call, the RN will ensure all lab results have been reviewed with the patient and discuss PrEP tolerability and adherence. At the 4-week follow-up, the RN will repeat steps in the initial visit, facilitate renewal of the electronic medication prescription, and review medication adherence.

At each follow-up visit, client's self-efficacy, attitudes/beliefs about PrEP, general health indicators, and social determinants of health, such as access to transportation and housing status, are recorded. Process evaluation will be performed to determine relationships of these variables and PrEP adherence, implementation (12 months), and continuation/dissemination (year 2) phases of the study. Outcome evaluation will occur after start-up and will include pre and post-enrollment rates of STI, rates of unplanned pregnancy, and post enrollment HIV seroconversion. The demographics characteristics of clients enrolled in the study will be compared to CANs existing PrEP populations served in traditional clinical settings. Qualitative information on barriers to PrEP initiation, barriers to adherence, and rationale for participation interruption/termination will be obtained by the PrEP nurses during monthly check-in appointments and telephone interviews. A portion of the study nurses' FTE will be dedicated to rapid analysis and reporting. This work will be managed in-kind by the Principal Investigator, Dr. Laura Armas-Kolostroubis, MD with 5% of FTE, with co-investigators Aleida Torres, DHSc., APRN with 30% FTE and Katy Wendel R.N., BSN with 15% FTE. Additional statistical analysis will be provided by Max Wilson, Ph.D. Final study publications will be completed by a panel of CAN stakeholders, including medical and prevention subject-matter experts (SMEs) and priority population members.

ELIGIBILITY:
Inclusion Criteria:

* Gay and bisexual men of color, cisgender women of color, and transgender women, transgender men, heterosexual men, Caucasian cisgender men and women individuals at risk for HIV and STI's, Individuals completing nPEP services. Between the ages of 18 and 65.

Exclusion Criteria:

* Minors younger than age 18, individuals not at risk for HIV, HIV positive status, HIV seroconversion, current or historical Hepatitis B virus infection, patients who are candidates for Truvada; patient has a history of renal dysfunction or eGFR values are below 60 mL/min, patients who are candidates for Descovy; patient has advanced CKD or an eGFR less than 30 mL/min, Patient is taking contraindicated medications*, patient has a positive pregnancy test or is breastfeeding. Any other clinical or psychosocial condition or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with dosing requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those who are aged 18-65 at the time of consent who are high risk patients for PrEP
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 | 18 months
  Demonstrate an increase of at least 10% (n=30) of target population members enrolled in pre-exposure prophylaxis services compared to baseline (n=300)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - CAN Community Health, Fort Lauderdale, Florida
  - CAN Community Health, Lake Worth, Florida
  - CAN Community Health, Miami Beach, Florida
  - CAN Community Health, Miami Gardens, Florida
  - CAN Community Health, Plantation, Florida

IPD SHARING:
Plan to Share IPD: No